CLINICAL TRIAL: NCT01913158
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter Study to Evaluate Safety and Efficacy of Anucort HC TM (Hydrocortisone Acetate) 25mg Rectal Suppositories in the Treatment of Symptomatic Internal Hemorrhoids
Brief Title: Safety and Efficacy Study of Anucort HC TM 25mg Rectal Suppositories to Treat Symptomatic Internal Hemorrhoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G & W Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRG-NY-13-002
Record Dates: First submitted 2013-05-24; First posted 2013-07-31 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Internal Hemorrhoids
MeSH Terms: interventions — Hydrocortisone; Suppositories

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo suppository (Placebo Comparator): Hydrogenated palm kernel oil suppositories
  Interventions: Drug: Placebo suppository
- Anucort-HC, 25 Mg Rectal Suppository (Active Comparator): Hydrocortisone Acetate suppositories
  Interventions: Drug: Anucort-HC, 25 Mg Rectal Suppository

INTERVENTIONS:
Drug: Anucort-HC, 25 Mg Rectal Suppository — Hydrocortisone acetate suppositories
  Other Names: Hydrocortisone acetate suppositories
  Arms: Anucort-HC, 25 Mg Rectal Suppository
Drug: Placebo suppository — Hydrogenated palm kernel oil suppositories
  Other Names: Hydrogenated palm kernel oil suppositories
  Arms: Placebo suppository

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of G&W Laboratories' Anucort HC TM (Hydrocortisone Acetate) 25mg Rectal Suppositories in subjects with internal hemorrhoidal symptoms.

DETAILED DESCRIPTION:
This is a randomized, vehicle-controlled, multicenter, double blind study of Anucort HC TM (Hydrocortisone Acetate) 25mg Rectal Suppositories in subjects with symptomatic internal hemorrhoids. Subjects will be randomly assigned in a 1:1 ratio to Test product or Vehicle, respectively.

Clinical evaluations will be performed at:

Visit 1/Day -3 (-1 day) to Day 1 Screening Visit 2/Day 1 Randomization (Start of Treatment) Visit 3/Day 8 (-1/+3 days) Interim Visit 4/Day 15 (-1/+3 days) End of Treatment / Early Termination Visit 5/ Day 28 (-1/+3 days)* 2 Weeks Post-Treatment/Follow-Up Phone Contact Safety will be assessed by monitoring adverse events (AEs) and clinically significant changes from Visit 1/Screening in laboratory values.

Number of Sites: Approximately 31 sites in the United States.

ELIGIBILITY:
Inclusion Criteria

1. Subjects with a diagnosis of symptomatic internal hemorrhoids will be selected to participate in the study.
2. Eligible subjects will be males or non-pregnant, non-lactating, non-menstruating females; ≥ 18 years of age; with diagnosis of Grade I, II or III internal hemorrhoidal disease.
3. For study entry the subject must have had anorectal bleeding during or after at least 2 of the 4 most recent attempted or successful bowel movements prior to Screening.
4. Subject may also have one or more other symptoms: pain, itching or throbbing.
5. At Visit 2/Day 1 (Randomization) subject must have recorded at least 2 instances of anorectal bleeding and no more than 1 incidence of no anorectal bleeding during attempted or successful bowel movements during the screening period between Visit 1/ Day -3 (Screening) and prior to Visit 2/Day 1 (Randomization).

Exclusion Criteria

1. History of permanent full-thickness rectal prolapse.
2. Current anal fissures and/or infective anal pathology.
3. Previous history of surgery for anorectal disease (within 1 year) or any other anorectal procedures
4. Subjects who are mentally incapacitated such that informed consent cannot be obtained.
5. Clinically significant co-morbid condition.
6. Diagnosis of Inflammatory Bowel Disease (IBD).
7. Evidence or history of fecal incontinence.
8. Clinically significant Laboratory values for hematology and chemistry .
9. Subjects who have had oral, transdermal, or injectable steroid therapy within days from Visit 1/Screening.
10. Presence of fissure or a fistula-in-ano, abscess, severe diverticular disease, polyps or colorectal adenoma or colorectal cancer, arteriovenous malformations, or any other pathological condition of the anus, colon or rectum other than symptomatic internal hemorrhoids which might be a potential cause of hematochezia.
11. Clinically significant systemic disease.
12. Pelvic radiation in the past or present.
13. Use of any venotropic medications within 7 days from Visit 2/Day 1.
14. Use of any anti-coagulant medications within 10 days from Visit 2/Day 1.
15. Use of topical/anorectal corticosteroids for hemorrhoidal therapy within 7 days from Visit 2/Day 1.
16. Use of topical/anorectal medicated hemorrhoidal therapy within 24 hours from Visit 2/Day 1.
17. Unable to cease use of OTC or prescription medications for treatment of hemorrhoidal disease during study period.
18. Immunocompromised subjects.
19. Known hypersensitivity or allergies to Hydrocortisone Acetate or any component of the IP (in any dosage form).
20. Use of any investigational drug or investigational device within 30 days prior to randomization.
21. Previous participation in this study.
22. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subjects ability to comply with study requirements.
23. Subjects unable to have a spontaneous bowl movement every day prior to randomization.
24. Rectal varicies or portal hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Bleeding Cessation | Up to 18 days
  The primary endpoint is bleeding cessation defined as cessation of anorectal bleeding associated with bowel movements or attempted bowel movements which does not recur after cessation for the remainder of the study period. The proportion of subjects with bleeding cessation using Anucort HCTM 25mg Rectal Suppositories will be compared statistically with the proportion of subjects using placebo.

SECONDARY OUTCOMES:
Improvement in the Severity Score of Pain | Up To 18 days
  Improvement in the Severity Score of Pain on the Visual Analogue Scale (VAS) from baseline to Visit 3/Day 8 and Visit 4 (End of Treatment)
Improvement in the Severity Score of Itching | Up to 18 days
  Improvement in the Severity Score of Itching from baseline to Visit 3/Day 8 and Visit 4 (End of Treatment)
Improvement in the Severity Score of Throbbing | Up to 18 days
  Improvement in the Severity Score of Throbbing to from baseline to Visit 3/Day 8 and Visit 4/Day 15 (End of Treatment)
Improvement in the Investigator Assessment | Up to 18 days
  Improvement in the Investigator Assessment
Improvement in the Subject Global Assessment | Up to 18 days
  Improvement in the Subject Global Assessment
Improvement in Severity of Bleeding | Up To 18 days
  Improvement in the severity of Bleeding from baseline to Visit 3/Day 8 and Visit 4 (End of Treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Allan G Coates, DO, Principal Investigator — Gastro Associates of Western Michigan
Locations (3):
- United States (3):
  - Clinical Research Associates, Huntsville, Alabama
  - IC Research, Sanford, Florida
  - Gastro Associates of Western Michigan, Wyoming, Michigan

IPD SHARING:
Plan to Share IPD: No